CLINICAL TRIAL: NCT02934113
Title: Worksite Interventions to Reduce Obesity and Diabetes Risk in Low SES Populations
Brief Title: "Working for You" Workplace Obesity Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201505131; R01DK103760 (NIH)
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Diabetes
Keywords: weight loss; text messaging; workplace; participatory approach; health care workers
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention)
- iOTA and HWPP (Experimental)
  Interventions: Behavioral: iOTA; Behavioral: HWPP
- HWPP (Experimental)
  Interventions: Behavioral: HWPP

INTERVENTIONS:
Behavioral: iOTA — The Individual Obesity Treatment Approach (iOTA) will assess individual behavior risks, collaborative goal-setting with a health coach, and the use of an interactive text system to provide ongoing support and self-monitoring of behavior change goals.
  Arms: iOTA and HWPP
Behavioral: HWPP — Work groups will participate in the Healthy Workplace Participatory Program (HWPP) to adapt and deploy interventions that change their work environments to support healthy eating and physical activity.
  Arms: HWPP; iOTA and HWPP

SUMMARY:
The purpose of this study is to test a workplace intervention program targeted at low SES workers. Working in partnership with BJC HealthCare, we will test an innovative multi-level intervention that includes an interactive obesity treatment program (iOTA) using SMS text messaging. The iOTA intervention will be embedded in a newly described Healthy Workplace Participatory Program, which incorporates employee participation in decision making to produce changes in the workplace environment that are acceptable, effective, and sustainable. These nested interventions will be tested a large delayed-start group-randomized trial. This study will rigorously test readily scalable interventions that can be translated to other work settings to reduce obesity and diabetes risk among low SES workers, a group at high risk for these disorders. This pragmatic clinical trial will advance the long-term goal of enabling employers and employees to reduce obesity and obesity-associated illnesses including diabetes.

DETAILED DESCRIPTION:
Specific Aim: Test a multi-level worksite weight loss intervention to help workers attain and maintain healthy weight. Investigators propose a new group-level participatory wellness program engaging all employees within intervention work groups. The proposed workplace participatory program will assist work groups to adapt and deploy interventions that change their work environments to support healthy eating and physical activity. Nested within this group-level intervention for all workers, obese (BMI>30) workers will be offered participation in an individual-level interactive obesity treatment approach (iOTA) intervention based on assessment of individual behavior risks, collaborative goal-setting with a health coach, and use of an interactive text system to provide ongoing support and self-monitoring of behavior change goals. Investigators will test these interventions in a delayed-start group randomized trial in 22 work groups (total workers = 990, obese workers = 308).

Specific Aim A: Implement and test a healthy workplace participatory program (HWPP) to promote healthy eating and healthy physical activity among all workers through changes in the work environment. Hypothesis: Workers in intervention groups will show improvements in healthy eating and activity compared to workers in control groups.

Specific Aim B: Implement and test an innovative Individual Obesity Treatment Approach (iOTA) in conjunction with changes in work environment. Hypothesis: Obese workers offered the iOTA intervention will lose weight over 24 month follow-up when compared to obese control group workers.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be a member of a chosen work group
* Speak English
* At least 18 years of age
* Sub-group (iOTA Intervention): BMI >=30, cell phone with text messaging capability

Exclusion Criteria:

* Sub-group (iOTA Intervention): pregnant or nursing, weight-loss surgery in past 12 mths, currently receiving chemotherapy or radiation treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1283 (Actual)
Dates: Start 2016-09; Primary Completion 2020-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Weight | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bradley A Evanoff, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will add data to the NIDDK data repository and share it in accordance with the NIDDK data sharing policy upon conclusion of the study.

REFERENCES:
- [Derived] Stein RI, Strickland JR, Tabak RG, Dale AM, Colditz GA, Evanoff BA. Design of a randomized trial testing a multi-level weight-control intervention to reduce obesity and related health conditions in low-income workers. Contemp Clin Trials. 2019 Apr;79:89-97. doi: 10.1016/j.cct.2019.01.011. Epub 2019 Jan 19. PMID 30664943
- [Derived] Tabak RG, Strickland JR, Stein RI, Dart H, Colditz GA, Kirk B, Dale AM, Evanoff BA. Development of a scalable weight loss intervention for low-income workers through adaptation of interactive obesity treatment approach (iOTA). BMC Public Health. 2018 Nov 16;18(1):1265. doi: 10.1186/s12889-018-6176-0. PMID 30445939